CLINICAL TRIAL: NCT05718024
Title: Impact of Night-time Dexmedetomidine-esketamine Infusion on Sleep Quality of Patients With Mechanical Ventilation or High-flow Nasal Cannula Oxygen Therapy in ICU: a Randomized Controlled Trial
Brief Title: Night-time Dexmedetomidine-esketamine Infusion and Sleep Quality in ICU Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Chief Physician, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-006
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Intensive Care Unit; Mechanical Ventilation; Dexmedetomidine; Esketamine; Sleep Quality
Keywords: Intensive care unit; Mechanical ventilation; Dexmedetomidine; Esketamine; Sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Analgesia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine-esketamine (Experimental): Dexmedetomidine-esketamine combination will be infused during night-time (8 pm to 6:30 am) for ICU patients with mechanical ventilation or high-flow nasal cannula oxygen therapy, for a duration of up to 5 days.
  Interventions: Drug: Dexmedetomidine-esketamine
- Control (Active Comparator): Propofol and remifentanil will be infused during night-time (8 pm to 6:30 am) for ICU patients with mechanical ventilation or high-flow nasal cannula oxygen therapy (if necessary), for a duration of up to 5 days.
  Interventions: Drug: Routine sedation and analgesia

INTERVENTIONS:
Drug: Dexmedetomidine-esketamine — Dexmedetomidine-esketamine combination will be infused during night-time (8 pm to 6:30 am) for ICU patients with mechanical ventilation or high-flow nasal cannula oxygen therapy.
  Arms: Dexmedetomidine-esketamine
Drug: Routine sedation and analgesia — Propofol and remifentanil will be infused during night-time (8 pm to 6:30 am) for ICU patients with mechanical ventilation or high-flow nasal cannula oxygen therapy (if necessary).
  Arms: Control

SUMMARY:
Dexmedetomidine and ketamine are both suggested for sedation and analgesia in ICU patients. Recent studies suggest that low-dose dexmedetomidine or ketamine/esketamine may improve sleep quality of ICU patients. The purpose of this trial is to observe whether night-time infusion of low-dose dexmedetomidine-esketamine combination can improve sleep structure of patients receiving mechanical ventilation or high-flow nasal cannula oxygen therapy in the ICU.

DETAILED DESCRIPTION:
Sleep disturbances are common in patients during intensive care unit (ICU) stay, especially those receiving mechanical ventilation. Persistent sleep disturbances are associated with negative outcomes, including increased sensitivity to pain, increased risk of delirium and cardiovascular events, and delayed weaning from mechanical ventilation.

Dexmedetomidine and ketamine are both suggested for sedation and analgesia in ICU patients. Previous studies showed that night-time dexmedetomidine infusion may improve sleep quality in ICU patients with mechanical ventilation, the effect is dose-dependent. However, sedative dose dexmedetomidine increases adverse events inculding bradycardia and hypotension. Recent studies suggest that ketamine/esketamine may also improve sleep quality. But even low-dose ketamine/esketamine increases adverse events including psychiatric and dissociative symptoms. We suppose that combined use of low-dose dexmedetomidine and esketamine may produce synergic effects in improving sleep quality in ICU patients with less adverse events.

The purpose of this trial is to observe whether night-time infusion of low-dose dexmedetomidine-esketamine combination can improve sleep structure of patients receiving mechanical ventilation or high-flow nasal cannula oxygen therapy in ICU patients and the safety of this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years or older;
* Admitted to the intensive care unit (ICU) after surgery;
* Receiving mechanical ventilation or high-flow nasal cannula oxygen therapy during night-time (after 6 pm), with an expected duration of ≥12 hours.

Exclusion Criteria:

* Duration of invasive/non-invasive ventilation ≥12 hours before enrollment;
* Planning to receive muscle relaxant treatment;
* History of schizophrenia, epilepsy, Parkinson's disease, or myasthenia gravis;
* Unable to communicate due to coma, delirium, severe dementia, or language barrier before receiving mechanical ventilation or high-flow nasal cannula oxygen therapy;
* Acute stroke or hypoxic encephalopathy, or after craniocerebral injury or neurosurgery;
* Comorbid with hyperthyroidism or pheochromocytoma;
* Taking sedative/hypnotic drugs or analgesics regularly (for more than 1 week) in the last month;
* LVEF<30%; sick sinus syndrome, severe sinus bradycardia (heart rate<50 beats/min), atrioventricular block of more than II degree and without pacemaker; or systolic blood pressure <90 mmHg despite vasopressor infusion;
* Severe liver dysfunction (Child-Pugh C grade), severe renal dysfunction (dialysis), or estimated survival ≤24 hours;
* Diagnosed obstructive sleep apnea, or body mass index >30 kg/m2;
* Allergies to dexmedetomidine and/or esketamine, or other conditions that are considered unsuitable for study participation;
* Enrolled in other clinical studies.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Percentage of non-rapid eye movement sleep stage 2 | From 21:00 pm to next 6:00 am during the first night after recruitment
  Polysomnographic monitoring is performed during the first night after recruitment with an EEG/PSG Recording System (SOMNO screen plus, SOMNO medics GmbH, Randersacker, Germany). The monitored sleep architecture is divided into wakefulness, non-rapid eye movement (stages N1, N2, and N3) sleep, and rapid eye movement (REM) sleep. The percentages of each sleep stage are calculated as the durations of each sleep stage divided by the total sleep time.

SECONDARY OUTCOMES:
Total sleep time | From 21:00 pm to next 6:00 am during the first night after enrollment
  Polysomnographic monitoring is performed during the first night after recruitment with an EEG/PSG Recording System (SOMNO screen plus, SOMNO medics GmbH, Randersacker, Germany). Total sleep time is defined as the summary of time spent in any sleep stage during the monitoring period.
Sleep efficiency | From 21:00 pm to next 6:00 am during the first night after enrollment
  Polysomnographic monitoring is performed during the first night after recruitment with an EEG/PSG Recording System (SOMNO screen plus, SOMNO medics GmbH, Randersacker, Germany). Sleep efficiency is calculated as the summary of time spent in each sleep stage divided by total sleep monitoring time.
Sleep fragmentation index | From 21:00 pm to next 6:00 am during the first night after enrollment
  Polysomnographic monitoring is performed during the first night after recruitment with an EEG/PSG Recording System (SOMNO screen plus, SOMNO medics GmbH, Randersacker, Germany). Sleep fragmentation index is calculated as the total number of awakenings and sleep-stage shifts divided by total sleep time.
Time of sleep in each stage | From 21:00 pm to next 6:00 am during the first night after enrollment
  Polysomnographic monitoring is performed during the first night after recruitment with an EEG/PSG Recording System (SOMNO screen plus, SOMNO medics GmbH, Randersacker, Germany). The monitored sleep architecture is divided into wakefulness, non-rapid eye movement (stages N1, N2, and N3) sleep, and rapid eye movement (REM) sleep.
Percentage of sleep in each stage (except percentage of non-rapid eye movement sleep stage 2) | From 21:00 pm to next 6:00 am during the first night after enrollment
  Polysomnographic monitoring is performed during the first night after recruitment with an EEG/PSG Recording System (SOMNO screen plus, SOMNO medics GmbH, Randersacker, Germany). The monitored sleep architecture is divided into wakefulness, non-rapid eye movement (stages N1, N2, and N3) sleep, and rapid eye movement (REM) sleep. The percentages of each sleep stage are calculated as the durations of each sleep stage divided by the total sleep time.
Pain intensity | During the first 5 days after enrollment
  Pain intensity is assessed twice daily (8:00 am to 10:00 am and 6:00 pm to 8:00 pm) with the numeric rating scale where 0=no pain and 10=the worst pain.
Subjective sleep quality | During the first 5 days after enrollment
  Subjective sleep quality is assessed daily (8:00 am to 10:00 am) with the numeric rating scale where 0=the best sleep and 10=the worst sleep.
Sedation-agitation level | During the first 5 days after enrollment
  Sedation-agitation level is assessed twice daily (8:00 am to 10:00 am and 6:00 pm to 8:00 pm) with the Richmond Agitation Sedation Scale; score ranges from -5 (unarousable) to +4 (combative) and 0 indicates alert and calm.
Delirium occurrence | During the first 5 days after enrollment
  Delirium is assessed twice daily (8:00 am to 10:00 am and 6:00 pm to 8:00 pm) with the Confusion Assessment Method for the ICU.
Duration of mechanical ventilation | Up to 30 days after enrollment
  Mechanical ventilation during ICU stay.
Length of ICU stay | Up to 30 days after enrollment
  Length of ICU stay.

OTHER OUTCOMES:
Length of hospital stay | Up to 30 days after enrollment
  Length of hospital stay.
Incidence of complications within 30 days | Up to 30 days after enrollment
  Complications are defined as new-onset medical conditions other than delirium that were deemed harmful and required therapeutic intervention, i.e., grade II or higher on the Clavien-Dindo classification.
All-cause mortality within 30 days | Up to 30 days after enrollment
  All-cause mortality within 30 days
Subjective sleep quality at 30 days | At 30 days after enrollment
  Subjective sleep quality is assessed with the Pittsburgh sleep quality index (PSQI). The PSQI consists of 19 self-rated and 5 other-rated items used to assess sleep quality over a month.
Quality of life at 30 days in physical domain | At 30 days after enrollment
  Quality of life is assessed with the World Health Organization Quality of Life-brief version (WHOQOL-BREF; a 24-item questionnaire that provides assessments of the quality of life in physical, psychological, and social relationship, and environmental domains. For each domain, the score ranges from 0 to 100, with higher score indicating better function).
Quality of life at 30 days in psychological domain | At 30 days after enrollment
  Quality of life is assessed with the World Health Organization Quality of Life-brief version (WHOQOL-BREF; a 24-item questionnaire that provides assessments of the quality of life in physical, psychological, and social relationship, and environmental domains. For each domain, the score ranges from 0 to 100, with higher score indicating better function).
Quality of life at 30 days in social relationship domain | At 30 days after enrollment
  Quality of life is assessed with the World Health Organization Quality of Life-brief version (WHOQOL-BREF; a 24-item questionnaire that provides assessments of the quality of life in physical, psychological, and social relationship, and environmental domains. For each domain, the score ranges from 0 to 100, with higher score indicating better function).
Quality of life at 30 days in environmental domain | At 30 days after enrollment
  Quality of life is assessed with the World Health Organization Quality of Life-brief version (WHOQOL-BREF; a 24-item questionnaire that provides assessments of the quality of life in physical, psychological, and social relationship, and environmental domains. For each domain, the score ranges from 0 to 100, with higher score indicating better function).

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friese RS. Sleep and recovery from critical illness and injury: a review of theory, current practice, and future directions. Crit Care Med. 2008 Mar;36(3):697-705. doi: 10.1097/CCM.0B013E3181643F29. PMID 18176314
- [Background] Elliott R, McKinley S, Cistulli P. The quality and duration of sleep in the intensive care setting: an integrative review. Int J Nurs Stud. 2011 Mar;48(3):384-400. doi: 10.1016/j.ijnurstu.2010.11.006. Epub 2010 Dec 24. PMID 21185560
- [Background] Parsons EC, Kross EK, Caldwell ES, Kapur VK, McCurry SM, Vitiello MV, Hough CL. Post-discharge insomnia symptoms are associated with quality of life impairment among survivors of acute lung injury. Sleep Med. 2012 Sep;13(8):1106-9. doi: 10.1016/j.sleep.2012.05.010. Epub 2012 Jul 2. PMID 22763017
- [Background] Combes A, Costa MA, Trouillet JL, Baudot J, Mokhtari M, Gibert C, Chastre J. Morbidity, mortality, and quality-of-life outcomes of patients requiring >or=14 days of mechanical ventilation. Crit Care Med. 2003 May;31(5):1373-81. doi: 10.1097/01.CCM.0000065188.87029.C3. PMID 12771605
- [Background] Granja C, Lopes A, Moreira S, Dias C, Costa-Pereira A, Carneiro A; JMIP Study Group. Patients' recollections of experiences in the intensive care unit may affect their quality of life. Crit Care. 2005 Apr;9(2):R96-109. doi: 10.1186/cc3026. Epub 2005 Jan 31. PMID 15774056
- [Background] Aurell J, Elmqvist D. Sleep in the surgical intensive care unit: continuous polygraphic recording of sleep in nine patients receiving postoperative care. Br Med J (Clin Res Ed). 1985 Apr 6;290(6474):1029-32. doi: 10.1136/bmj.290.6474.1029. PMID 3921096
- [Background] Friese RS, Diaz-Arrastia R, McBride D, Frankel H, Gentilello LM. Quantity and quality of sleep in the surgical intensive care unit: are our patients sleeping? J Trauma. 2007 Dec;63(6):1210-4. doi: 10.1097/TA.0b013e31815b83d7. PMID 18212640
- [Background] Gehlbach BK, Chapotot F, Leproult R, Whitmore H, Poston J, Pohlman M, Miller A, Pohlman AS, Nedeltcheva A, Jacobsen JH, Hall JB, Van Cauter E. Temporal disorganization of circadian rhythmicity and sleep-wake regulation in mechanically ventilated patients receiving continuous intravenous sedation. Sleep. 2012 Aug 1;35(8):1105-14. doi: 10.5665/sleep.1998. PMID 22851806
- [Background] Elliott R, McKinley S, Cistulli P, Fien M. Characterisation of sleep in intensive care using 24-hour polysomnography: an observational study. Crit Care. 2013 Mar 18;17(2):R46. doi: 10.1186/cc12565. PMID 23506782
- [Background] Slatore CG, Goy ER, O'hearn DJ, Boudreau EA, O'Malley JP, Peters D, Ganzini L. Sleep quality and its association with delirium among veterans enrolled in hospice. Am J Geriatr Psychiatry. 2012 Apr;20(4):317-26. doi: 10.1097/JGP.0b013e3182487680. PMID 22367162
- [Background] Finan PH, Goodin BR, Smith MT. The association of sleep and pain: an update and a path forward. J Pain. 2013 Dec;14(12):1539-52. doi: 10.1016/j.jpain.2013.08.007. PMID 24290442
- [Background] Fernandes NM, Nield LE, Popel N, Cantor WJ, Plante S, Goldman L, Prabhakar M, Manlhiot C, McCrindle BW, Miner SE. Symptoms of disturbed sleep predict major adverse cardiac events after percutaneous coronary intervention. Can J Cardiol. 2014 Jan;30(1):118-24. doi: 10.1016/j.cjca.2013.07.009. Epub 2013 Oct 16. PMID 24140074
- [Background] Kjolhede P, Langstrom P, Nilsson P, Wodlin NB, Nilsson L. The impact of quality of sleep on recovery from fast-track abdominal hysterectomy. J Clin Sleep Med. 2012 Aug 15;8(4):395-402. doi: 10.5664/jcsm.2032. PMID 22893770
- [Background] Kanji S, Mera A, Hutton B, Burry L, Rosenberg E, MacDonald E, Luks V. Pharmacological interventions to improve sleep in hospitalised adults: a systematic review. BMJ Open. 2016 Jul 29;6(7):e012108. doi: 10.1136/bmjopen-2016-012108. PMID 27473952
- [Background] Stanchina ML, Abu-Hijleh M, Chaudhry BK, Carlisle CC, Millman RP. The influence of white noise on sleep in subjects exposed to ICU noise. Sleep Med. 2005 Sep;6(5):423-8. doi: 10.1016/j.sleep.2004.12.004. Epub 2005 Mar 31. PMID 16139772
- [Background] Freedman NS, Gazendam J, Levan L, Pack AI, Schwab RJ. Abnormal sleep/wake cycles and the effect of environmental noise on sleep disruption in the intensive care unit. Am J Respir Crit Care Med. 2001 Feb;163(2):451-7. doi: 10.1164/ajrccm.163.2.9912128. PMID 11179121
- [Background] Parthasarathy S, Tobin MJ. Effect of ventilator mode on sleep quality in critically ill patients. Am J Respir Crit Care Med. 2002 Dec 1;166(11):1423-9. doi: 10.1164/rccm.200209-999OC. Epub 2002 Sep 5. PMID 12406837
- [Background] Cooper AB, Thornley KS, Young GB, Slutsky AS, Stewart TE, Hanly PJ. Sleep in critically ill patients requiring mechanical ventilation. Chest. 2000 Mar;117(3):809-18. doi: 10.1378/chest.117.3.809. PMID 10713011
- [Background] Fanfulla F, Ceriana P, D'Artavilla Lupo N, Trentin R, Frigerio F, Nava S. Sleep disturbances in patients admitted to a step-down unit after ICU discharge: the role of mechanical ventilation. Sleep. 2011 Mar 1;34(3):355-62. doi: 10.1093/sleep/34.3.355. PMID 21358853
- [Background] Trompeo AC, Vidi Y, Locane MD, Braghiroli A, Mascia L, Bosma K, Ranieri VM. Sleep disturbances in the critically ill patients: role of delirium and sedative agents. Minerva Anestesiol. 2011 Jun;77(6):604-12. PMID 21617624
- [Background] Weinhouse GL, Watson PL. Sedation and sleep disturbances in the ICU. Crit Care Clin. 2009 Jul;25(3):539-49, ix. doi: 10.1016/j.ccc.2009.04.003. PMID 19576529
- [Background] Gabor JY, Cooper AB, Crombach SA, Lee B, Kadikar N, Bettger HE, Hanly PJ. Contribution of the intensive care unit environment to sleep disruption in mechanically ventilated patients and healthy subjects. Am J Respir Crit Care Med. 2003 Mar 1;167(5):708-15. doi: 10.1164/rccm.2201090. PMID 12598213
- [Background] Schiza SE, Simantirakis E, Bouloukaki I, Mermigkis C, Arfanakis D, Chrysostomakis S, Chlouverakis G, Kallergis EM, Vardas P, Siafakas NM. Sleep patterns in patients with acute coronary syndromes. Sleep Med. 2010 Feb;11(2):149-53. doi: 10.1016/j.sleep.2009.07.016. Epub 2010 Jan 18. PMID 20083431
- [Background] Nelson LE, Lu J, Guo T, Saper CB, Franks NP, Maze M. The alpha2-adrenoceptor agonist dexmedetomidine converges on an endogenous sleep-promoting pathway to exert its sedative effects. Anesthesiology. 2003 Feb;98(2):428-36. doi: 10.1097/00000542-200302000-00024. PMID 12552203
- [Background] Alexopoulou C, Kondili E, Diamantaki E, Psarologakis C, Kokkini S, Bolaki M, Georgopoulos D. Effects of dexmedetomidine on sleep quality in critically ill patients: a pilot study. Anesthesiology. 2014 Oct;121(4):801-7. doi: 10.1097/ALN.0000000000000361. PMID 24988068
- [Background] Xia ZQ, Chen SQ, Yao X, Xie CB, Wen SH, Liu KX. Clinical benefits of dexmedetomidine versus propofol in adult intensive care unit patients: a meta-analysis of randomized clinical trials. J Surg Res. 2013 Dec;185(2):833-43. doi: 10.1016/j.jss.2013.06.062. Epub 2013 Jul 24. PMID 23910886
- [Background] Wu XH, Cui F, Zhang C, Meng ZT, Wang DX, Ma J, Wang GF, Zhu SN, Ma D. Low-dose Dexmedetomidine Improves Sleep Quality Pattern in Elderly Patients after Noncardiac Surgery in the Intensive Care Unit: A Pilot Randomized Controlled Trial. Anesthesiology. 2016 Nov;125(5):979-991. doi: 10.1097/ALN.0000000000001325. PMID 27571256
- [Background] Sun YM, Zhu SN, Zhang C, Li SL, Wang DX. Effect of low-dose dexmedetomidine on sleep quality in postoperative patients with mechanical ventilation in the intensive care unit: A pilot randomized trial. Front Med (Lausanne). 2022 Aug 31;9:931084. doi: 10.3389/fmed.2022.931084. eCollection 2022. PMID 36117973
- [Background] Barrett W, Buxhoeveden M, Dhillon S. Ketamine: a versatile tool for anesthesia and analgesia. Curr Opin Anaesthesiol. 2020 Oct;33(5):633-638. doi: 10.1097/ACO.0000000000000916. PMID 32826629
- [Background] Kaur U, Pathak BK, Singh A, Chakrabarti SS. Esketamine: a glimmer of hope in treatment-resistant depression. Eur Arch Psychiatry Clin Neurosci. 2021 Apr;271(3):417-429. doi: 10.1007/s00406-019-01084-z. Epub 2019 Nov 19. PMID 31745646
- [Background] Song B, Zhu J. A Novel Application of Ketamine for Improving Perioperative Sleep Disturbances. Nat Sci Sleep. 2021 Dec 25;13:2251-2266. doi: 10.2147/NSS.S341161. eCollection 2021. PMID 34992482
- [Background] Feinberg I, Campbell IG. Ketamine administration during waking increases delta EEG intensity in rat sleep. Neuropsychopharmacology. 1993 Aug;9(1):41-8. doi: 10.1038/npp.1993.41. PMID 8397722
- [Background] Ahnaou A, Huysmans H, Biermans R, Manyakov NV, Drinkenburg WHIM. Ketamine: differential neurophysiological dynamics in functional networks in the rat brain. Transl Psychiatry. 2017 Sep 19;7(9):e1237. doi: 10.1038/tp.2017.198. PMID 28926001
- [Background] Duncan WC, Sarasso S, Ferrarelli F, Selter J, Riedner BA, Hejazi NS, Yuan P, Brutsche N, Manji HK, Tononi G, Zarate CA. Concomitant BDNF and sleep slow wave changes indicate ketamine-induced plasticity in major depressive disorder. Int J Neuropsychopharmacol. 2013 Mar;16(2):301-11. doi: 10.1017/S1461145712000545. Epub 2012 Jun 7. PMID 22676966
- [Background] Faraguna U, Vyazovskiy VV, Nelson AB, Tononi G, Cirelli C. A causal role for brain-derived neurotrophic factor in the homeostatic regulation of sleep. J Neurosci. 2008 Apr 9;28(15):4088-95. doi: 10.1523/JNEUROSCI.5510-07.2008. PMID 18400908
- [Background] Bunney BG, Li JZ, Walsh DM, Stein R, Vawter MP, Cartagena P, Barchas JD, Schatzberg AF, Myers RM, Watson SJ, Akil H, Bunney WE. Circadian dysregulation of clock genes: clues to rapid treatments in major depressive disorder. Mol Psychiatry. 2015 Feb;20(1):48-55. doi: 10.1038/mp.2014.138. Epub 2014 Nov 4. PMID 25349171
- [Background] Bartova L, Papageorgiou K, Milenkovic I, Dold M, Weidenauer A, Willeit M, Winkler D, Kasper S. Rapid antidepressant effect of S-ketamine in schizophrenia. Eur Neuropsychopharmacol. 2018 Aug;28(8):980-982. doi: 10.1016/j.euroneuro.2018.05.007. Epub 2018 Jul 2. PMID 30041987
- [Background] Molero P, Ramos-Quiroga JA, Martin-Santos R, Calvo-Sanchez E, Gutierrez-Rojas L, Meana JJ. Antidepressant Efficacy and Tolerability of Ketamine and Esketamine: A Critical Review. CNS Drugs. 2018 May;32(5):411-420. doi: 10.1007/s40263-018-0519-3. PMID 29736744
- [Background] Canuso CM, Singh JB, Fedgchin M, Alphs L, Lane R, Lim P, Pinter C, Hough D, Sanacora G, Manji H, Drevets WC. Efficacy and Safety of Intranasal Esketamine for the Rapid Reduction of Symptoms of Depression and Suicidality in Patients at Imminent Risk for Suicide: Results of a Double-Blind, Randomized, Placebo-Controlled Study. Focus (Am Psychiatr Publ). 2019 Jan;17(1):55-65. doi: 10.1176/appi.focus.17105. Epub 2019 Jan 7. PMID 32015715
- [Background] Segmiller F, Ruther T, Linhardt A, Padberg F, Berger M, Pogarell O, Moller HJ, Kohler C, Schule C. Repeated S-ketamine infusions in therapy resistant depression: a case series. J Clin Pharmacol. 2013 Sep;53(9):996-8. doi: 10.1002/jcph.122. Epub 2013 Jul 24. No abstract available. PMID 23893490
- [Background] Persson J, Hasselstrom J, Maurset A, Oye I, Svensson JO, Almqvist O, Scheinin H, Gustafsson LL, Almqvist O. Pharmacokinetics and non-analgesic effects of S- and R-ketamines in healthy volunteers with normal and reduced metabolic capacity. Eur J Clin Pharmacol. 2002 Feb;57(12):869-75. doi: 10.1007/s002280100353. PMID 11936706
- [Background] Bornemann-Cimenti H, Wejbora M, Michaeli K, Edler A, Sandner-Kiesling A. The effects of minimal-dose versus low-dose S-ketamine on opioid consumption, hyperalgesia, and postoperative delirium: a triple-blinded, randomized, active- and placebo-controlled clinical trial. Minerva Anestesiol. 2016 Oct;82(10):1069-1076. Epub 2016 Jun 21. PMID 27327855
- [Background] Hu ZC, Xu G, Zhang XW, Ma K, Jin JJ, Li PS. [Meta-analysis of the effects of dexmedetomidine combined with ketamine during dressing changes in burn patients]. Zhonghua Shao Shang Za Zhi. 2020 Jun 20;36(6):458-464. doi: 10.3760/cma.j.cn501120-20190327-00145. Chinese. PMID 32594705
- [Background] Lee KH, Lee SJ, Park JH, Kim SH, Lee H, Oh DS, Kim YH, Park YH, Kim H, Lee SE. Analgesia for spinal anesthesia positioning in elderly patients with proximal femoral fractures: Dexmedetomidine-ketamine versus dexmedetomidine-fentanyl. Medicine (Baltimore). 2020 May;99(20):e20001. doi: 10.1097/MD.0000000000020001. PMID 32443302
- [Background] Austin PC. An Introduction to Propensity Score Methods for Reducing the Effects of Confounding in Observational Studies. Multivariate Behav Res. 2011 May;46(3):399-424. doi: 10.1080/00273171.2011.568786. Epub 2011 Jun 8. PMID 21818162